CLINICAL TRIAL: NCT05385939
Title: Impact of Transition to a New Single Patient Room NICU on Gastric Bacterial Colonization of Preterm Neonates Compared to a Traditional Open Bay NICU
Brief Title: Gastric Bacterial Colonization of Preterm Neonates
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Other Study IDs: Christiana Care Health System
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Microbial Colonization; Preterm Birth
MeSH Terms: conditions — Communicable Diseases; Premature Birth | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Time period 1: Time period one included infants admitted to the current traditional, open bay NICU.
  Interventions: Other: Observational
- Time period 2: Time period 2 included infants admitted to the private, single family room NICU.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This was an observational study which involved collection of stool samples and environmental samples at 1 week and 4 weeks of life.

SUMMARY:
This prospective cohort study was conducted in the Christiana Care Health System Neonatal Intensive Care Unit. It occurred at two time periods: Time period 1 included infants admitted to the traditional, open bay NICU. Time period 2 included infants admitted to the new private, single family room NICU. There was a 3 month period between Time period 1 and Time period 2 to ensure that there was no patient overlap. Stool samples and environmental samples were collected at 1 and 4 weeks after birth in both time periods. The objective of this study was to establish the gastrointestinal microbiome of infants born at less than 32 weeks gestation admitted to the exiting open bay NICU and compare it to the gastrointestinal microbiome of infants born at less than 32 weeks admitted to the new private, single family room NICU.

ELIGIBILITY:
Inclusion Criteria:

* Less than 32 weeks gestation at birth

Exclusion Criteria:

* Infants in Time period 2 that were admitted to the traditional, open bay NICU

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of infants born at less than 32 weeks born and admitted to the CCHS NICU. Infants in Time period 2 that were admitted to the traditional, open bay NICU will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Microorganisms identified in stool samples | 4 weeks
  Microorganisms identified in stool samples obtained at weeks 1 and 4 of life using the 16s rRNA sequencing based technique.

SECONDARY OUTCOMES:
Microorganisms identified in environmental samples | 4 weeks
  Microorganisms identified in samples obtained from the counter, floor, and incubator top or inside wall at weeks 1 and 4 of life using the 16 s rRNA sequencing based technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Christiana Care Health Services, Inc., Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No